CLINICAL TRIAL: NCT07398534
Title: PICO Negative Pressure for the Treatment of Uninfected Foot Ulcers and Wound Dehiscence - an Unblinded, Randomized-controlled, Superiority Trial (BALPIC Trial)
Brief Title: PICO Negative Pressure for Uninfected Foot Ulcers and Wound Dehiscence (BALPIC)
Acronym: BALPIC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ilker Uckay (Other)
Responsible Party: Sponsor-Investigator, Ilker Uckay, Prof. Dr. med. Ilker Uçkay, Balgrist University Hospital
Organization: Balgrist University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BASEC 2025-D0043
Record Dates: First submitted 2026-01-29; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Wound Dehiscence; Wound
Keywords: acute wound; negative pressure vacuum therapy; prospective-randomized trial
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: Unblinded, prospective-randomized superiority trial in favor of PICO use
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PICO (Experimental): Application of PICO 7 Single Use NPWT System at -80 mmHg for a minimum of 7 days. PICO therapy may be continued for up to 42 days based on clinical necessity. Device change every 7 days. Wound assessment weekly. SMITH & NEPHEW MEDICAL LTD. PICO 7 15CM X 20CM; NEGATIVE PRESSURE WOUND THERAPY POWERED SUCTION PUMP (UDI 04582111156419). The PICO system creates a closed environment over the wound, evacuating exudate into an absorptive dressing while promoting wound closure through controlled suction.
  Interventions: Procedure: Professional Wound Care
- Professional Wound CAre (Other): Professional wound debridement by specialized wound nurses, including dressing changes and local antiseptics if clinically indicated, without the use of any negative pressure device. Treatment for up to 42 days based on clinical necessity. Wound assessment weekly. Individualized professional wound care according to hospital and Swiss nursing guidelines. The intensity of debridement, dressing type, and antiseptic use lies at the discretion of the wound nurse and will be recorded.
  Interventions: Procedure: Professional Wound Care

INTERVENTIONS:
Procedure: Professional Wound Care — Professional wound debridement by specialized wound nurses, including dressing changes and local antiseptics if clinically indicated, without the use of any negative pressure device. Treatment for up to 42 days based on clinical necessity. Wound assessment weekly.
  Individualized professional wound care according to hospital and Swiss nursing guidelines. The intensity of debridement, dressing type, and antiseptic use lies at the discretion of the wound nurse and will be recorded.

SUMMARY:
The investigators compare negative pressure wound therapy (NPWT) using the PICO 7 system versus professional wound debridement alone in adult orthopedic patients with acute, non-infected wound dehiscence or diabetic foot ulcers. Patients are randomized 1:1 to either PICO therapy (minimum 7 days, up to 42 days) or standard wound care (professional debridement without NPWT). The primary outcome is wound closure without surgical revision at Day 42. The trial is stratified for diabetic foot ulcers to enable subgroup analysis.

DETAILED DESCRIPTION:
Acute postoperative wound dehiscence and foot ulcers represent a frequent clinical challenge in adult orthopedic patients worldwide. According to institutional data, wound dehiscence occurs in 2-5% of elective orthopedic procedures, depending on surgery type, patient comorbidities, and obesity. Among patients with diabetes, approximately half will develop foot ulcers during their lifetime.

The management of non-infected wounds can be either surgical (revision surgery with primary closure) or conservative (professional debridement and wound care with or without negative pressure wound therapy). Despite widespread clinical experience with NPWT in orthopedic surgery, high-quality prospective evidence remains scarce. The orthopedic literature lacks adequately powered randomized controlled trials comparing NPWT to standard wound care for acute, non-infected wound dehiscence.

The investigators hypothesize that NPWT leads to superior wound closure rates (85% vs. 70%) and accelerated healing compared to professional debridement alone. The PICO Single Use Negative Pressure Wound Therapy System creates a closed environment over the wound, evacuating exudate into an absorptive dressing while promoting secondary closure through controlled suction at -80 mmHg.

The BALPIC trial evaluates a therapeutic concept rather than comparing different NPWT devices. Infected wounds are excluded, as NPWT is conventionally avoided over purulent wounds to allow free drainage. Wound assessment is performed by specialized wound nurses using standardized measurements and photographic documentation.

ELIGIBILITY:
Inclusion Criteria:

* - Age ≥ 18 years
* Able to consent
* Patient of orthopaedic surgery or of the (Diabetic) Foot Polyclinic at the Balgrist University Hospital
* Presence of an acute, dehiscent, clinically uninfected wound requiring additional measures
* First episode of wound treatment for the actual wound (no recurrences) in the last 12 months
* Wound measuring ≥ 0.5 cm in wide, length or depth
* 42 days of scheduled follow-up
* Bacterial orthopaedic infections of any nature, independently of implants or co-morbidities; according to clinical, laboratory, radiological, microbiological features of infection
* First or second episode of infection

Exclusion Criteria:

* - Patient's individual refusal to participate
* Patient already treated with any vacuum-assisted wound device for any wound in the last 12 months; independently of therapy success, the hospital or the localization of the prior wound
* Underlying liquor leak (spine surgery)
* Visually active bleeding from the wound
* Wound size >10 cm in any dimension
* Anticipated active clinical follow-up of less than 42 days
* Other wound treatments besides PICO and debridement (e.g. hyperbaric oxygen therapy, other negative-pressure devices, local antibiotics, local antibiotic dressings) (however, local antiseptics and dressing changes remain allowed)
* Immediate surgical wound revision in the operating theatre for closure
* Planned plastic or reconstructive surgery already at inclusion

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-01-29 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Wound closure without surgical revision at Day 42 | Day 42 (±7 days)
  Wound closure is defined as reduction of wound size by a minimum of 90% compared to baseline, without need for surgical revision. Wound failure is defined as persistent wound (less than 90% reduction) after 42 days or surgical wound revision during the study period.

SECONDARY OUTCOMES:
2. Rapidity of wound closure | Day 7, 14, 21, 28, 35, and 42
  Time to achieve 90% wound size reduction.
Wound closure without surgical revision at Day 7, 14, 21, 28, and 35 | Day 7, 14, 21, 28, and 35 (±2 days)
  Binary assessment of wound closure at each weekly visit
4. Wound closure for diabetic foot ulcers only (stratified analysis) | Day 42 (±7 days)
  Pre-specified subgroup analysis for DFU patients.
5. Adverse events related to wound therapy | Day 1 to Day 42 (±7 days)
  All adverse events during the therapy and follow-up time, including device deficiencies in the PICO arm.
6. Length of hospital stay | Day 1 to Day 42 (±7 days)
  Duration of hospital stay in acute care setting.
7. Overall costs of hospitalization | Day 1 to Day 42 (±7 days)
  Total hospitalization costs.

CONTACTS AND LOCATIONS:
Overall Officials: Ilker Uçkay, Prof. Dr. med., Principal Investigator — Balgrist University Hospital, University of Zurich, Zurich, Swizerland
Locations (1):
- Balgrist University Hospital, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
The investigators may share anonymized key elements upon reasonable scientific request to the corresponding persons
Supporting Information: Study Protocol, ICF, CSR
Time Frame: After the final analysis
Access Criteria: Reasonable scientific request to the corresponding Sponsor-Investigator
URL: https://www.balgrist.ch/